CLINICAL TRIAL: NCT07265921
Title: A Phase I First-in-Human, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0609 in Adult Participants With Locally Advanced/Metastatic Solid Tumors
Brief Title: A Phase I Study of SIM0609 in Adult Participants With Locally Advanced/Metastatic Solid Tumors
Acronym: Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianwei Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0609-101
Record Dates: First submitted 2025-11-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Cancer
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A dose escalation of SIM0609 (Experimental): Multiple dose levels of SIM0609 will be explored in dose escalation, and determine the maximum tolerated dose.
  Interventions: Drug: SIM0609 for injection
- A dose expansion of SIM0609 -CRC cohort (Experimental): 1~3 dose levels of SIM0609 will be explored in dose expansion to evaluate the preliminary anti-tumor activity of SIM0609 in colorectal carcinoma (CRC)
  Interventions: Drug: dose expansion of SIM0609 in CRC
- A dose expansion of SIM0609-GC/GEJC cohort (Experimental): 1~3 dose levels of SIM0609 will be explored in dose expansion to evaluate the preliminary anti-tumor activity of SIM0609 in gastric/gastroesophageal junction adenocarcinoma (GC/GEJC)
  Interventions: Drug: dose expansion of SIM0609 in GC/GEJC cohort
- A dose expansion of SIM0609-PDAC cohort (Experimental): 1~3 dose levels of SIM0609 will be explored in dose expansion to evaluate the preliminary anti-tumor activity of SIM0609 in pancreatic ductal adenocarcinoma (PDAC)
  Interventions: Drug: dose expansion of SIM0609 in PDAC cohort
- A dose expansion of SIM0609-positive other solid tumors cohort (Experimental): 1~3 dose levels of SIM0609 will be explored in dose expansion to evaluate the preliminary anti-tumor activity of SIM0609 in positive other solid tumors
  Interventions: Drug: dose expansion of SIM0609 in positive other solid tumors

INTERVENTIONS:
Drug: SIM0609 for injection — Multiple dose levels of SIM0609 will be explored in dose escalation
  Arms: A dose escalation of SIM0609
Drug: dose expansion of SIM0609 in CRC — 1~3 dose levels of SIM0609 will be explored in dose expansion to evaluate the preliminary anti-tumor activity of SIM0609 in colorectal carcinoma (CRC)
  Arms: A dose expansion of SIM0609 -CRC cohort
Drug: dose expansion of SIM0609 in GC/GEJC cohort — 1~3 dose levels of SIM0609 will be explored in dose expansion in GC/GEJC cohort
  Arms: A dose expansion of SIM0609-GC/GEJC cohort
Drug: dose expansion of SIM0609 in PDAC cohort — 1~3 dose levels of SIM0609 will be explored in dose expansion in PDAC cohort
  Arms: A dose expansion of SIM0609-PDAC cohort
Drug: dose expansion of SIM0609 in positive other solid tumors — 1~3 dose levels of SIM0609 will be explored in positive other solid tumors cohort
  Arms: A dose expansion of SIM0609-positive other solid tumors cohort

SUMMARY:
This is an open-label,multicenter phase I study to evaluate the safety,Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of SIM0609 in Adult Participants with Locally Advanced/Metastatic Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signature of informed consent form;
2. At least 18 years old, male or female;
3. Participants with histologically and/or cytologically confirmed locally advanced/metastatic solid tumors;
4. Participants should have at least one evaluable or measurable tumor lesion;
5. Participants have failed the standard of therapy in the locally advanced/metastatic setting;
6. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1;
7. Expected survival ≥12 weeks;
8. Adequate organ and bone marrow function;
9. Availability of archival formalin-fixed, paraffin-embedded (FFPE) tumor tissue, or fresh biopsies within 28 days before first administration, is mandatory

Exclusion Criteria:

1. Active second primary malignancies within the previous 2 years except for localized cancers that are considered to have been cured and in the opinion of the Investigator present a low risk for recurrence;
2. Symptomatic central nervous system (CNS) metastases or CNS metastases requiring CNS-directed local therapy or corticosteroid treatment that occurred within 2 weeks prior to the first administration of the investigational treatment;
3. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging screening;
4. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study ;
5. Any active infections requiring systemic therapy within 2 weeks prior to the initiation of the study treatment;
6. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring drainage or medical intervention within 4 weeks before the first dose of study treatment;
7. Not recovered from previous anticancer therapy-induced AEs(Adverse Events);
8. Currently participating or has participated in a study of an investigational agent or using an investigational device within 4 weeks of first dose of study treatment;
9. Received prior therapies within the following time frames prior to the first dose of study treatment:

   1. Previous cytotoxic therapy, anticancer targeted small molecules within 2 weeks.
   2. Anti-cancer antibody, immune checkpoint inhibitor or ADC within 5 half-lives or 4 weeks (whichever is shorter).
   3. Chinese medicines/herbal preparations with anticancer indication taken within 2 weeks.
   4. Radiation therapy within 4 weeks.
10. Prior exposure to topoisomerase I inhibitor (TOP1i)-based antibody drug conjugate (ADC) therapies or CDH17-targeted ADC therapies.
11. Use of any live vaccine therapy within 4 weeks prior to the first dose of study treatment.
12. Administration of below medications ≤14 days prior to the first dose of study treatment.

    1. Strong or moderate CYP3A4 inducers/inhibitors;
    2. Drugs with known risk of Torsades de Pointes(TdP);
    3. Drugs that may prolong the QT interval;
13. Major surgery within 2 weeks of receiving the first dose of study treatment;
14. Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome ;
15. Active or chronic hepatitis B or hepatitis C infection;
16. Participants with clinically significant cardiovascular diseases;
17. History of allogeneic organ transplantation or graft-versus-host disease;
18. History of hypersensitivity to active or inactive excipients of SIM0609 or drugs with a similar chemical structure or class to SIM0609;
19. Pregnant or nursing (lactating) women;
20. Male participants with female partners of reproductive potential, unless they are using highly effective contraceptive methods from signing of informed consent to 180 days after the last dose of study treatment;
21. Presence of any other condition that may increase the risk associate with study participant or may interfere with the interpretation of study results, and, in the opinion of the Investigator, would make the participant inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Dose escalation:Dose -limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 21/28days)
Dose escalation:Safety and Tolerability | 2 years
  Safety and tolerability: Incidence and severity of AEs and serious adverse events (SAEs) assessed by CTCAE v5.0, changes in laboratory values, vital signs, and ECGs. AE related dose interruptions, dose reduction and treatment discontinuation, dose intensity
Dose escalation: Objective response rate(ORR) | 2 years
  Proportion of subjects who have a complete or partial response assessed by investigator per RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing
  - Jiangsu Province Hospital, Nanjing
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital，Fudan University, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No